CLINICAL TRIAL: NCT04315519
Title: Investigation of the Effect of Blood Flow Restricted Aerobic Exercise on Cardiorespiratory Fitness and Blood Glucose in Type 2 Diabetes Mellitus
Brief Title: Effect of Blood Flow Restricted Aerobic Exercise in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Elif ŞAHİN, Principal investigator, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26
Record Dates: First submitted 2020-01-27; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
Keywords: Blood Flow Restricted Exercise; Type 2 Diabetes; Aerobic Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restricted Aerobic (BFRA) (Experimental): Low intensity Aerobic exercise with Blood Flow Restriction
  Interventions: Other: Exercise
- Moderate Aerobic Exercise (MAE) (Experimental): moderate intensity aerobic exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Aerobic Exercise

SUMMARY:
Comparison of the effect of low intensity blood flow restricted aerobic exercise on glycemic and respiratory status with moderate aerobic exercise.

DETAILED DESCRIPTION:
The aim of this study is to show, whether the effect of low-intensity aerobic exercise training combined with blood flow restriction is similar on both glycemic and cardiorespiratory status compared to moderate-intensity continuous aerobic exercise, in individuals with "type 2 diabetes mellitus" .

ELIGIBILITY:
Inclusion Criteria:

* Having Type 2 Diabetes
* Not have been recruited any exercise programme for 6 months
* Volunteering to participate in the study

Exclusion Criteria:

* Nephropathy
* Retinopathy
* Have had myocardial infarction at least 6 months ago
* Stable or unstable angina pectoris
* The presence of peripheral artery disease
* Resting blood pressure above 160/100 mmHg
* Body mass index over 35 kg / m2
* History of deep vein thrombosis, pulmonary embolism or stroke

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | up to 12 months
  Fasting Blood Glucose, this data will be collected from the individulas routine biochemistry tests
HbA1c | up to 12 months
  Glycated hemoglobin, This data will be collected from teh individulas during routine test
Blood Glucose in Oral glucose Tolerance Test | Up to 12 months
  Blood Glucose in Oral glucose Tolerance Test, this data will be collected from the individuals during routine tests.
Cardiorespiratory Fitness | Up to 12 months
  Maximal Power in Maximal Exercise Test, this test will be performed in incremental cardiopulmonary exercise test in cycle ergometer.

SECONDARY OUTCOMES:
The Strength of Quadriceps Muscle | Up to 12 months
  The Strength of Quadriceps Muscle, this data will be collected before the intervention eith a manual muscle tester, in sitting position.
Fat Free Mass | Up to 12 months
  Fat Free Mass will be calculated by bioimpedance analysis, this data will be collected with all individulas to see the changes with the muscle mass, the test will be The test will be carried out with a 4-channel test device, both hand and foot, to eveluate changes segmentally.
The Strength of Hamstring Muscle | Up to 12 months
  The Strength of Hamstring Muscle, this data will be collected before the intervention eith a manual muscle tester, in sitting position.

IPD SHARING:
Plan to Share IPD: Undecided